CLINICAL TRIAL: NCT03413800
Title: A Phase II, Open-label Study of Lenalidomide and Dexamethasone Followed by Donor Lymphocyte Infusions in Relapsed Multiple Myeloma Following Allogeneic Stem Cell Transplant
Brief Title: Len/Dex/DLI in Relapsed Multiple Myeloma After Allogeneic Stem Cell Transplant
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: Celgene (Industry); C3i Center Inc. (Unknown)
Responsible Party: Principal Investigator, Jean Roy, MD, Ciusss de L'Est de l'Île de Montréal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMR003
Record Dates: First submitted 2018-01-15; First posted 2018-01-29 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Relapsed Hematologic Malignancy; Multiple Myeloma
Keywords: hematopoietic stem cell transplant; lenalidomide; DLI
MeSH Terms: conditions — Hematologic Neoplasms; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Lenalidomide-Dexamethasone-DLI (Experimental): 1. Patients will receive Len (10 mg in the presence of ≤ grade I acute GVHD or absence of chronic GVHD; 5 mg in presence of controlled mild or moderate chronic GVHD) daily x 21 days with Dex 40 mg once weekly for a total of 6 cycles of 28 days each
     1. For grade ≥III non hematologic or grade IV hematologic toxicity, Len can be reduced to 5 mg
     2. In absence of these toxicities, acute GVHD (using Glucksberg modified criteria) or severe chronic GVHD (using NIH criteria), Len dose can be increased by 5 mg per cycle to a maximum of 25 mg
  2. If eligibility is confirmed, sibling and unrelated donor transplant recipients will both receive 3 donor lymphocyte infusions (DLIs) at the following doses: 5 x 106 CD3+/kg; 1 x 107 CD3+/kg; 5 x 107 CD3+/kg
  3. Patient will be followed for 5 years post relapse.
  Interventions: Drug: Lenalidomide-Dexamethasone-DLI

INTERVENTIONS:
Drug: Lenalidomide-Dexamethasone-DLI — Lenalidomide (Len) and Dexamethasone (Dex) for 6 months followed by three donor lymphocyte infusions (DLIs)

SUMMARY:
Multiple Myeloma (MM) is a morbid disease which can only be cured with an allogeneic hematopoietic stem cell transplant (HSCT). Approximately 50% of allotransplanted patients will relapse, with a median survival of 5 years. Better approaches to improve disease control at relapse, while decreasing toxicity, are urgently needed.

Relapse after allogeneic transplant is a failure of the graft versus MM effect (GvMM). DLIs can be used to control disease following relapse, but the optimal dose, schedule of administration and drug association remain elusive, while the immunosuppression found in MM patients can compromise their effect. One reason for immunotherapy failure relates to the immunological environment: as much as myeloma cells depend on their microenvironment to survive and proliferate, the immunotherapeutic effect of allogeneic HSCT depends on both systemic and local immunological status to be efficacious. Immunomodulatory drugs such as Lenalidomide (Len) have been tried in various settings after allogeneic transplantation with the aim to reverse immunosuppression and stimulate the GvMM, but if and how Len influences a GvMM and thereby promotes an immunotherapeutic success remained uncharacterized. Therefore, a deeper understanding of the immunological environment in MM patients is needed in order to establish and / or restore a potent GvMM effect.

This study proposes the powerful combination of the two following goals, one clinical and one biological :

1. Clinical: The investigators propose a two-step treatment using first Len in association with Dexamethasone (Dex), followed by Donor Leukocytes Infusions (DLIs) to offer an optimal disease control strategy in relapsed patients. The cytoreductive and immunomodulatory effects of Len is expected to induce a permissive immunological environment for the immunotherapeutic activity of DLIs to develop, while the association with Dex will lessen the risk of graft-versus-host disease (GVHD). This treatment combination has the potential to further improve depth of myeloma response, delay myeloma progression and improve patient survival.
2. Biological: In an attempt to gain knowledge on how the GvMM behaves in MM patients post-relapse after having received a combined treatment of Len/Dex/DLIs, the investigators propose to characterize the immune environment of their bone marrow (BM) using both minimal residual disease (MRD) assessement by flow cytometry and an unbiased analysis of the transcriptome at various time points.

DETAILED DESCRIPTION:
Myeloma patients in first relapse after sibling or unrelated donor allogeneic transplant willing to participate in this study will be screened for eligibility.

1. After baseline evaluation including BM aspirate for plasma cell count, minimal residual disease using 8-color multiparameter flow cytometry, transcriptome sequencing and a positron emission tomography (PET scan), patients will receive Len- Dex daily x 21 days with Dex 40 mg once weekly for a total of 6 cycles of 28 days each
2. Patients will then be evaluated clinically for acute and chronic GVHD before each cycle and a PET scan will be performed at the end of Len/Dex treatment
3. Sibling and unrelated donor transplant recipients will receive 3 DLIs
4. Disease and immune evaluation using serum and urine electrophoresis/immunofixation in addition to measurement of serum-free light chains, BM aspirate for plasma cell count and minimal residual disease using 8-color multiparameter flow cytometry, transcriptome sequencing and a PET scan will be performed

   1. A BM aspirate will be performed before each DLI for plasma cell count, MRD evaluation by flow cytometry and transcriptome sequencing
   2. Patients will be followed with a BM aspirate every 3 months x 1 year, then yearly and at progression for plasma cell count and evaluation
   3. Transcriptome sequencing will be done on BM aspirates at time of relapse, after Len/Dex cycles, 6m, 12m, 18m and 24m after the last-DLI.
   4. A PET scan will be performed after the last DLI and at progression.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years
2. Myeloma patients in first relapse after a sibling or unrelated allogeneic stem cell transplantation
3. Patients with measurable disease at time of relapse based on the IMWG criteria
4. All study participants must comply with the Revlimid Pregnancy Prevention Plan.
5. Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid Pregnancy Prevention Plan.

   Exclusion Criteria:
6. Relapse occurred within 180 days post allograft
7. Refractory to Len at any given time before allogeneic transplantation
8. Presence of ≥ grade II or uncontrolled acute GVHD
9. Presence of severe or uncontrolled chronic GVHD
10. Karnofsky score < 70%
11. Bilirubin > 50 μmol/L unless felt to be related to Gilbert's disease or hemolysis; AST and ALT > 5 x upper limit of normal (ULN); alkaline phosphatase > 5 x ULN
12. Known hypersensitivity to Len or Dex
13. Active infection with any of the following viruses: HIV, HTLV-1 or 2, hepatitis B (defined as HBsAg positivity) or hepatitis C (defined as anti-HCV positivity or HCV-RNA positivity)
14. Presence of another malignancy with an expected survival estimated < 75% at 5 years (complete resection of basal cell carcinoma or squamous cell carcinoma, complete resection of a ductal carcinoma in situ, presence of lobular carcinoma in situ, complete resection of carcinoma in situ of the cervix, or an in situ or low-risk prostate cancer after curative therapy are not exclusion criteria)
15. Positive beta-human chorionic gonadotropin pregnancy test, to be performed in all women of childbearing potential at screening and baseline. Female study participants who are surgically sterile (hysterectomy) or who have been postmenopausal for at least 12 consecutive months are automatically eligible for this criterion
16. Females of child-bearing potential not agreeing to remain abstinent or to use 2 simultaneous effective methods of contraception from at least 4 weeks before, to at least 4 weeks following discontinuation of Len. Males not agreeing to use a condom during any sexual contact with females of child-bearing potential from at least 4 weeks before, to at least 4 weeks following discontinuation of Len
17. Women who are lactating
18. Female of child-bearing potential who are planning to become pregnant while enrolled in this study up to 4 weeks after the last Len dose
19. Participation in a trial with an investigational agent within 30 days prior to entry in the study
20. Inability to provide written informed consent prior to initiation of any study-related procedures, or inability, in the opinion of investigators, to comply with all requirements of the study
21. Estimated probability to survive less than 6 months after initiation of Len and Dex
22. Current history of drug and/or alcohol abuse
23. Any abnormal condition or laboratory result that is considered by investigators capable of altering patient's condition, compliance or study outcome
24. Any patient who, in the opinion of investigators, should not participate in this study
25. Having received allogeneic stem cell transplantation in relapse after autologous transplant.
26. Having received Len therapy after allogeneic transplant, before relapse
27. Poor organ function defined as either: diffusing capacity of the lung for carbon monoxide corrected for hemoglobin using Dinakara method (DLCOc) < 50%; forced expiratory volume in 1 second < 50%; left ventricular ejection fraction (LVEF) < 40% evaluated by echocardiogram or multi-gated acquisition scan (MUGA); uncontrolled arrhythmia; symptomatic cardiac disease; creatinine clearance < 30 mL/minute; liver cirrhosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Len-Dex-DLI in patients with relapsed myeloma measured by progression-free survival | 2 years
  To determine the as efficacy of Len and Dex followed by DLIs, measured by progression-free survival at 2 years after the last DLI

SECONDARY OUTCOMES:
Incidence of grade ≥III non hematologic toxicity and incidence of grade ≥IV hematologic toxicity | 5 years
  Patients will be evaluated according to protocol and adverse events will be monitored continuously, documented and collected in database
Incidence of acute GVHD | 1 years
  GVHD will be evaluated according to protocol, documented and collected in database. Analysis will be done by cumulative incidence.
Incidence of chronic GVHD | 2 years
  GVHD will be evaluated according to protocol, documented and collected in database. Analysis will be done by cumulative incidence.
Maximum grades of acute and chronic GVHD | 2 years
  GVHD will be evaluated according to protocol, documented and collected in database
Response to treatment | 3 years
  International Myeloma Working Group (IMWG) response after Len/Dex and after DLIs, best response achieved
Non-relapse mortality after DLIs | 3 years
  Analysis by cumulative incidence
Overall survival at 2 years | 2 years
  Kaplan Meier analysis
Incidence of progression at 2 years | 2 years
  Kaplan Meier analysis
Disease status assessment by flow cytometry | 5 years
  BM evaluation of minimal residual disease (MRD) by multiparametric flow cytometry (MFC) analysis
Disease status assessment by PET scan | 5 years
  Evaluation of extramedullary disease by positron emission tomography (PET) scan
Evaluation of quality of life (QoL) during treatment | 5 years
  QoL questionnaire will be given to patients according to protocol
Evaluation of the BM microenvironment by transcriptome analysis before and after treatments | 3 years
  Both mononucleated celles and extracellular compartment will be analyzed by RNAseq

CONTACTS AND LOCATIONS:
Overall Officials: Jean Roy, MD, Principal Investigator — Ciusss de L'Est de l'Île de Montréal
Locations (1):
- CIUSSS de l'Est-de-l'île-de-Montréal, Installation Hôpital Maisonneuve Rosemond, Montreal, Quebec, Canada